CLINICAL TRIAL: NCT00974844
Title: Posterior Assisted Levitation by Pars-Plana Levitator
Brief Title: Posterior Assisted Levitation of Dropped Nucleus
Acronym: PAL
Status: Completed | Type: Observational
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jamshed Ahmed, Assistant Professor, Dow University of Health Sciences
Other Study IDs: DUHS-SWJA
Record Dates: First submitted 2009-08-24; First posted 2009-09-10 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2009-09

CONDITIONS: Cataract
Keywords: posterior assisted levitation; Pars Plana; Dropped nucleus; cataract; complication of; surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Dropping of nucleus is a common complication during cataract extraction by phacoemulsification. The investigators describe a new technique to retrieve the dropped nucleus by using an instrument called Pars Plana Levitator (ASICO-LLC, USA).

DETAILED DESCRIPTION:
Upon recognition of posterior capsular rupture and dropping of nucleus phaco prob will be withdrawn, status of the nucleus will be visualized by posterior segment non contact lens and if the nucleus found floating, pars plana levitator will be introduced through temporal pars plana, its prongs will be opened and nucleus will be grasped between prongs. Nucleus will be lifted up till the anterior chamber where phacoemulsification will be performed in a usual manner and a posterior chamber intraocular lens will be implanted if possible in the remaining bag.

ELIGIBILITY:
Inclusion Criteria:

* Patients during cataract surgery whose nucleus will be dropped during phacoemulsification

Exclusion Criteria:

* Completely dropped nucleus touching the posterior pole

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had dropped nucleus during phacoemulsification
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Wahab, FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Eye Unit III, Lyari General Hospital , Dow university of Health Sciences, Karachi, Sindh, Pakistan